CLINICAL TRIAL: NCT05340426
Title: Porcine Kidney Xenotransplantation in Patients With End-Stage Kidney Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Approval to move forward with this clinical trial has not been granted by governing bodies.
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: United Therapeutics (Industry); Lung Biotechnology PBC (Industry)
Responsible Party: Principal Investigator, Jayme E Locke, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300008933
Record Dates: First submitted 2022-02-27; First posted 2022-04-22 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Kidney Failure, Chronic
Keywords: Pig Kidney; Porcine Kidney; End Stage Kidney Disease; UKidney
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Transplantation, Heterologous

STUDY DESIGN:
Intervention Model Description: Phase I clinical trial involving the use of a porcine kidney xenograft for transplant in place of a human kidney allograft to treat chronic renal failure in patients on dialysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Porcine Kidney (UKidney) transplant (Experimental): In this phase I single arm study patients with acute renal failure will be transplanted with a porcine xenograft versus a human allograft-after transplantation the best practice standard of care will be followed for monitoring and immunosuppression with the exception of additional monitoring for potential porcine transmitted infections
  Interventions: Device: UKidney

INTERVENTIONS:
Device: UKidney — The intended clinical product is a kidney derived from a domestic pig that contains an intentional genomic alteration (IGA) to protect it after transplantation from the human immune response via inactivation of endogenous porcine genes responsible for expression of pig epitopes and inclusion of human transgenes to inhibit host immunogenic response.
  Other Names: Porcine Kidney; Xenotransplant

SUMMARY:
The mismatch between organ supply and demand results in the deaths of thousands of Americans each year. Our research group aims to solve this unmitigated health care crisis by translating advances in xenotransplantation to humans and expanding organ supply in a sustainable fashion using genetically modified pigs as a source of organs. We propose here a phase I clinical trial of porcine kidney xenotransplantation into 20 people with end-stage kidney disease. Source donor animals are pigs with 10 gene edits (10-GE) which attenuate immunologic harm to the kidney xenograft. 10-GE pigs are housed in a designated pathogen-free facility within 30 minutes of the transplantation center. Xenotransplantation procedures follow conventional practices currently employed in allotransplantation and comply with multiple regulatory standards to ensure ethical treatment of research subjects and source animals. Recruitment and xenotransplantation will occur over 5 years with study follow-up extending 1 year after xenotransplantation. Primary outcome variables surround patient safety, such as patient survival and the rate of zoonotic disease transmission. Secondary outcome variables include commonly used metrics of graft survival and function.

DETAILED DESCRIPTION:
Twenty patients with ESKD listed for kidney allotransplantation at UAB will be enrolled to receive either one or two porcine kidney xenotransplants from a 10-GE pig donor, contingent on the pig's overall size at the time of procurement.

Recruitment and xenotransplantation will occur over a five-year time period. Patients will undergo follow-up of one year post-xenotransplant with study extension if graft survival exceeds one year.

Participants will undergo prospective crossmatching with a 10-GE pig to determine histocompatibility prior to xenotransplant. After performance of a negative crossmatch, procurement of the donor pig will occur in a surgical suite at the designated pathogen-free facility near the UAB campus where the donor herd is maintained.

Porcine kidney(s) will be transported under sterile and hypothermic conditions to the main UAB hospital. The porcine kidney(s) will be transplanted into the research subject in standard surgical fashion within the abdomen and immunosuppression will be administered. The induction immunosuppression regimen utilized will mirror that used in human-to-human allotransplantation; this regimen represents current standard-of-care. After transplantation, kidney health will be assessed biochemically, histologically, and radiographically. Subjects will be monitored for potential zoonotic disease transmission and blood-based chimerism as well as thrombocytopenia or indicators of consumptive coagulopathy, development of anti-human leukocyte antigen antibody/alloantibody sensitization.

FOLLOW-UP PHASE

Xenotransplant recipients are expected to remain in the hospital under close clinical surveillance by the study team and associates for approximately 1-3 weeks, pending kidney recovery and surveillance for potential complications.

Post-transplant Medications. The post-transplant immunosuppression and maintenance regimen consists of conventional agents that are routinely used in kidney allotransplantation. Although immunosuppression practices in allotransplantation can vary widely from center to center, the approach below utilizes agents and doses employed by UAB's Incompatible Kidney Transplant Program. As the ideal immunosuppression regimen for xenotransplantation has not yet been established, Investigator and team have adopted strategies used in incompatible kidney allotransplantation based on the assumption that significant antigenic variation remains between the species and antibody responses of unknown specificity below the level of detection of the crossmatch may impact later function or graft longevity.

Maintenance immunosuppression will be administered as below:

Note: Induction immunosuppression will be given at the time of xenotransplantation and will include ATG 1.5mg/kg, solumedrol 500mg, and eculizumab 1200mg. The remaining doses of ATG will be given to a total of 6mg/kg to complete induction. The ATG dosing schedule will vary depending on degree of hemolysis and/or lineage depletion, as is routinely done in allotransplantation.

Tacrolimus in divided doses daily, to a target level of 8-12 ng/mL Mycophenolate Mofetil (1000mg twice daily as a starting dose and tapered as needed per UAB incompatible kidney allotransplantation protocol) Daily prednisone, tapered from induction to a target dose of 10 mg per day. Eculizumab, 1200 mg every two weeks Investigator and study team have opted to include eculizumab as a maintenance agent to avert or attenuate complement-mediated injury of the graft. Although the 10-GE pig expresses a number of human transgenes designed to regulate complement biology, the finding of TMA in the brain-dead human recipient (*Porrett et al, AJT 2022) suggests that additional blockade of complement may be beneficial. Given that eculizumab increases the risk of infection with encapsulated bacteria, research subjects will be required to complete the FDA REMS and be vaccinated accordingly. Ciprofloxacin 500 mg twice daily (adjusted for GFR) for 6 weeks after transplantation in individuals vaccinated with meningococcal vaccine as above. Subjects will be monitored and counseled about side effects of prolonged ciprofloxacin use, such as tendonitis and tendon rupture. When eculizumab is discontinued (such as after graft removal), ciprofloxacin will be discontinued 6 weeks after the last eculizumab dose.

Thrombosis Prophylaxis: Recipients may be maintained on a heparin infusion and/or receive aspirin as clinically indicated. Subcutaneous heparin will be administered for DVT prophylaxis. Early ambulation will be encouraged.

Antimicrobial Prophylaxis: Surgical wound prophylaxis will be discontinued within 24h of exiting the operating room. Prophylaxis against opportunistic infections will be continued after transplant.

For PCP prophylaxis: Sulfamethoxazole (or Dapsone if allergic to Sulfa). This will be continued for 12 months.

For viral/CMV/HSV prophylaxis:

Valganciclovir to prevent CMV reactivation if recipient is CMV positive. This will be renally dosed and continued for 6 months post-transplant.

If recipient is CMV negative, valacylovir will be selected for HSV prophylaxis and continued for 6 months post-transplant.

Note: Although the transplantation of CMV+ donors to CMV- recipients occurs often in human allotransplantation, this situation is unlikely to occur in the setting of this trial as porcine donors in the DPF are CMV negative. Should a porcine donor test positive for CMV, prophylaxis in the recipient would be altered accordingly (i.e., valganciclovir or ganciclovir would be provided in consultation with Transplant Infectious Disease specialists)

For Candidal prophylaxis (i.e. oral thrush): Nystatin swish/swallow

Follow-up Visits and Procedures

Frequency:

Xenotransplant recipients will be closely monitored for the duration of their participation in the study. After discharge from the hospital, the study team anticipates seeing these patients in the outpatient clinic according to the table below, with additional clinic visits as needed. Recipients will have 24h access to the study team and will be extensively educated about clinical triggers (i.e., signs and symptoms of infection, myocardial infarction, etc.) to seek care. Each visit will consist of routine care for kidney transplant patients, including an assessment of medication compliance, collection of vital signs, history, a review of systems, and physical examination including examination of the surgical wound (for the first 6-8 weeks after transplantation

Post-transplant time period Clinic visit schedule 0-1 months Twice Weekly 2-3 months Weekly 3-6 months Twice Monthly 6-12 months (or study endpoint) Monthly

Protocol biopsies will occur 24h after transplant, 3 months, 6 months, and at 12 months assuming graft survival. Biopsies may be performed either percutaneously or may require an open surgical approach. Percutaneous biopsies will be performed under ultrasound guidance. Biopsy schedule may be amended for cause. Biopsies will be submitted for routine pathologic analysis (H&E, immunofluorescence microscopy, etc.), as well as research studies. Biopsy findings will be scored using the Banff criteria.

Imaging Studies:

Ultrasound: Kidney xenograft perfusion will be monitored with ultrasound. Grafts will be studied with ultrasound daily for the first week then weekly thereafter while recipients are in the hospital. Monthly ultrasounds will be performed in the outpatient setting for the first year (or for the duration of the graft if less than one year). Schedule may be amended for cause.

Nuclear medicine scanning: Kidney perfusion scans will be performed monthly to acquire additional information about xenograft excretion and perfusion.

Laboratory Assessments:

Most of the laboratory tests below will be performed daily for the first 2 weeks after transplantation and then gradually transition to weekly and/or monthly schedules pending clinical stability of the recipient. Testing schedule may be escalated for cause. Tests will be performed on either blood or urine and are largely non-invasive or minimally invasive (such as phlebotomy). This testing schedule will largely replicate the routine monitoring of transplant recipients.

Complete blood count with differential Complete metabolic panel (including LFTs) Coagulation panel (including PT/PTT/INR) Tacrolimus level Mycophenolate level Urinalysis Urine culture 24h urine collection (Creatinine, Protein, Albumin, Urea, Sodium, Potassium, Protein Electrophoresis and Immunofixation etc.) Daily on postoperative day 1,2,3 Weekly for two weeks Monthly for first year Random urine protein Random urine creatinine Vit D 25 and Vit D 1,25 level Intact PTH Hemoglobin A1C Lipid Profile Lymphocyte profiling (e.g. CD4, CD8,CD19, CD20) Note: blood will also be analyzed in the research laboratory where higher dimensional immune profiling can be performed using multiparameter flow cytometry, single-cell RNA-sequencing, etc.) Iron, TIBC, Ferritin Samples for blood chimerism studies Immunologic monitoring Single antigen bead screening to assess for changes in anti-HLA antibody titers which may have been provoked by cross-reactivity with SLA.

Retrospective crossmatch Pathogen monitoring CMV PCR will be performed monthly for the first transplant year. Serum and urine will be tested monthly for BK virus reactivation for one year. Monitoring of donor-derived infection

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75 years
* Body mass index (BMI) 18-40 kg/m2
* Waitlisted for kidney allotransplantation at UAB
* Dialysis dependent
* Proficient in the English language
* Presence of risk factors for

  * high wait list mortality, AND/OR
  * anticipated or actual prolonged wait time on the wait list, AND/OR
  * inability to access a suitable organ offer.
  * Note: Examples of risk factors include high cPRA, frequent incompatible crossmatches leading to prolonged wait times, listing at an advanced age, and impending loss of dialysis access, recurrent disease in previous transplants.
* Crossmatch compatible with porcine donor
* SARS-CoV-2 vaccination in accordance with most recent CDC guidance
* Willingness to obtain other standard-of-care vaccinations for kidney transplant recipients (MMR, HBV, Herpes Zoster, etc.) and for patients receiving eculizumab (Menactra® and Bexsero®)
* Reside within a 60-minute radius of the UAB hospital (by ground transport)

Exclusion Criteria:

* Age <18y or ≥ 76y
* BMI ≤ 18 or ≥ 41 kg/m2
* Current pregnancy
* Presence of severe comorbid disease, including but not limited to uncontrolled HTN or DM (hemoglobin A1C (HgA1C) >10%), advanced cardiovascular disease, absent surgical targets for implantation, etc.
* Presence of hypercoagulable disorder
* Inability to accept a blood transfusion
* Intolerance of immunosuppression
* History of medical non-compliance
* Presence of untreated psychiatric disease
* Significant psychosocial vulnerability and/or poor social support
* Current use/abuse of illicit drugs and/or abuse of alcohol
* History of psychiatric hospitalization
* Inability to provide informed consent
* Pre-emptive transplant
* Inability to comply with study protocols and procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient Survival After Porcine Transplant | 30 days
  These time points align with both biologic events that occur after transplantation (i.e., immune reconstitution after T cell depletion) as well as conventional transplant outcome metrics used by regulatory authorities (i.e., Organ Procurement and Transplantation Network, United Network for Organ Sharing)
Patient Survival After Porcine Transplant | 90 days
  These time points align with both biologic events that occur after transplantation (i.e., immune reconstitution after T cell depletion) as well as conventional transplant outcome metrics used by regulatory authorities (i.e., Organ Procurement and Transplantation Network, United Network for Organ Sharing)
Patient Survival After Porcine Transplant | 6 months
  These time points align with both biologic events that occur after transplantation (i.e., immune reconstitution after T cell depletion) as well as conventional transplant outcome metrics used by regulatory authorities (i.e., Organ Procurement and Transplantation Network, United Network for Organ Sharing)
Patient Survival After Porcine Transplant | 12 months
  These time points align with both biologic events that occur after transplantation (i.e., immune reconstitution after T cell depletion) as well as conventional transplant outcome metrics used by regulatory authorities (i.e., Organ Procurement and Transplantation Network, United Network for Organ Sharing)
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Post-op day 1
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Post-op day 2
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Post-op day 3
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Week 1
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Week 2
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Month 1
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Month 2
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Month 3
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Month 4
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Month 5
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Month 6
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Month 7
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Month 8
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Month 9
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Month 10
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Month 11
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of thrombocytopenia or indicators of consumptive coagulopathy after transplant with porcine kidney | Month 12
  Consumptive coagulopathy has been observed in some non-human primate models of transplant with a pig kidney. Thrombocytopenia was also observed in the UAB brain-dead recipient but could not be attributed to the porcine kidney given the altered physiology of brain death.
Prevalence of blood based chimerism after transplantation | Post-op day 1
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Post-op day 2
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Post-op day 3
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Week 1
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Week 2
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Month 1
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Month 2
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Month 3
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Month 4
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Month 5
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Month 6
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Month 7
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Month 8
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Month 9
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Month 10
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Month 11
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Prevalence of blood based chimerism after transplantation | Month 12
  The presence of donor-derived cells in the blood stream of a transplant recipient can either portend graft versus host disease (GVHD) or be diagnostic of the disease
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Post-op day 1
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Post-op day 2
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Post-op day 3
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Week 1
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Week 2
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Month 1
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Month 2
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Month 3
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Month 4
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Month 5
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Month 6
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Month 7
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Month 8
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Month 9
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Month 10
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Month 11
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.
Development of anti-human leukocyte antigen (HLA) antibody/alloantibody sensitization after transplant with a porcine kidney | Month 12
  It is currently unknown whether porcine kidney xenografts will ever function sufficiently to become a destination therapy for patients with ESKD. However, if porcine kidney xenografts have modest longevity, there may be benefit to temporary rescue from dialysis. Porcine kidney xenografts may then act as a bridge to human allotransplantation. Thus, there is the need to determine whether porcine kidney xenografts provoke the development of anti-HLA antibody and sensitize recipients against human allografts. Such sensitization may prevent xenograft recipients from ever receiving a human allotransplant, and the frequency of this event must be determined in order to counsel patients effectively about the risks of participating in additional trials of xenotransplantation.

SECONDARY OUTCOMES:
Kidney outcomes including: | Through study completion, an average of 1 year
  • Dialysis-free survival-patient remains off of dialysis
Kidney outcomes including: | Through study completion, an average of 1 year
  • estimated glomerular filtration rate (eGFR)
Kidney outcomes including: | Through study completion, an average of 1 year
  • urine output during index hospitalization
Kidney outcomes including: | Through study completion, an average of 1 year
  • prevalence and degree of proteinuria
Kidney outcomes including: | Through study completion, an average of 1 year
  • incidence and duration of delayed graft function (DGF)
  o DGF defined as need for at least one dialysis session in first week after transplantation
Kidney outcomes including: | Through study completion, an average of 1 year
  • incidence of primary non-function (PNF)
  o PNF defined as dialysis dependence or creatinine clearance ≤ 20 ml/min 90 days after transplantation
Histologic outcomes including: | Through study completion, an average of one year
  * incidence of acute cellular rejection (ACR)
  * incidence of antibody-mediated rejection (AMR)
  * incidence of complement deposition, etc.
  * incidence of recurrent disease
Infectious outcomes including: | Through study completion, an average of one year
  * incidence of surgical site infections
  * incidence of hospital acquired infection (i.e. pneumonia, urinary tract infection (UTI), Central Line-Associated Blood Stream Infection (CLABSI))
  * prevalence of conventional opportunistic infection (i.e. pneumocystis pneumonia (PCP), cytomegalovirus (CMV), polyomavirus (BK) etc.);
Immunologic outcomes: | Through study completion, an average of one year
  • calculated panel reactive antibody (cPRA)
Cardiovascular outcomes including: | Through study completion, an average of one year
  • resolution or exacerbation of hypertension (HTN), ease of blood pressure control as evidenced by type and number of anti-hypertensive medications
Cardiovascular outcomes including: | Through study completion, an average of one year
  • rate of new onset diabetes after transplant (NODAT) or worsening/improvement of control of pre-existing diabetes mellitus (DM) as evidenced by medications needed for glycemic control
Cardiovascular outcomes including: | Through study completion, an average of one year
  • incidence of myocardial infarction and/or stroke following xenotransplantation
Cardiovascular outcomes including: | Through study completion, an average of one year
  • incidence of hypotension or other blood pressure alterations, as renin produced by the pig kidney may not be able to cleave human angiotensinogen, evidenced by type and dosage of anti-hypertensive or anti-hypotensive medications required to maintain blood pressure within normal limits of 160/80

CONTACTS AND LOCATIONS:
Overall Officials: Jayme E Locke, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bobier C, Reinhardt N, Pawlowski K. Animal rights, animal research, and the need to reimagine science. New Bioeth. 2024 Mar;30(1):63-76. doi: 10.1080/20502877.2023.2300232. Epub 2024 Jan 5. PMID 38182130